CLINICAL TRIAL: NCT00379509
Title: Phase I Radiosensitization Study of GW572016 With Biologic Correlates in Locoregionally Recurrent Breast Cancer
Brief Title: Lapatinib and Radiation Therapy in Treating Patients With Locally Recurrent or Chemotherapy-Refractory Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0411; P30CA016086 (NIH)
Record Dates: First submitted 2006-09-20; First posted 2006-09-22 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — Lapatinib; Gene Expression Profiling; Microarray Analysis; Immunohistochemistry; Biopsy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GW572016 (Experimental)
  Interventions: Drug: lapatinib ditosylate; Genetic: TdT-mediated dUTP nick end labeling assay; Genetic: gene expression analysis; Genetic: microarray analysis; Other: immunohistochemistry staining method; Procedure: biopsy; Radiation: radiation therapy

INTERVENTIONS:
Drug: lapatinib ditosylate — Patients will be assigned in cohorts of 3. Dose levels of GW572106 will include 500mg, 1000mg,1500 mg (additional levels at 750 mg and 1250 mg will be added if needed). Lapatinib is an oral drug. It is taken every day.
Genetic: TdT-mediated dUTP nick end labeling assay — Genetic analysis of tumor tissue
Genetic: gene expression analysis — Genetic analysis of tumor tissue.
Genetic: microarray analysis — Genetic analysis of tumor tissue.
Other: immunohistochemistry staining method — Laboratory analysis of tumor tissue.
Procedure: biopsy — Serial biopsies by skin punch or core biopsy or fine needle aspiration.
Radiation: radiation therapy — Radiotherapy will be delivered at standard dose and fractionation. For patients who have not received previous locoregional radiotherapy, 50-56 Gy will be delivered to the regional lymph nodes and/or chest wall at a dose of 2 Gy per fraction, 5 days per week followed by a boost to the sites of gross involvement to a total dose of 60-70 Gy over a course of 6-7 weeks. For patients who have received adjuvant radiotherapy, a dose of 35-45 Gy will be delivered to sites of chest wall involvement at a dose of 1.8 Gy per fraction over 4-5 weeks. In either de novo or reirradiated settings, the total dose to the brachial plexus will not exceed 60 Gy.

SUMMARY:
RATIONALE: Lapatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving lapatinib together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of lapatinib when given together with radiation therapy in treating patients with locally recurrent or chemotherapy-refractory locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity of lapatinib ditosylate and radiotherapy in patients with locally recurrent breast cancer or chemotherapy-refractory, locally advanced or metastatic breast cancer.
* Determine the impact of this drug on inhibition of receptor and downstream signal transduction pathway activation in tumor tissue, in the context of inhibitor dose escalation with or without radiotherapy.

Secondary

* Determine, preliminarily, the efficacy of lapatinib ditosylate and radiotherapy in these patients.
* Correlate response in these patients with inhibition of downstream signaling.
* Assess gene expression changes in tumor biopsy samples from patients treated with lapatinib ditosylate alone or in combination with radiotherapy.

OUTLINE: This is a multicenter, parallel group, dose-escalation study of lapatinib ditosylate. Patients are stratified according to prior radiotherapy (yes vs no).

* Group I (prior radiotherapy): Patients receive oral lapatinib ditosylate once daily in the absence of disease progression or unacceptable toxicity. Beginning on day 8 of lapatinib ditosylate therapy, patients undergo concurrent radiotherapy 5 days a week for up to 5 weeks.
* Group II (no prior radiotherapy): Patients receive oral lapatinib ditosylate as in group I. Beginning on day 8, patients undergo concurrent radiotherapy 5 days a week for up to 7 weeks.

In each group, cohorts of 3-6 patients receive escalating doses of lapatinib ditosylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during the first course.

Patients undergo skin punch or core biopsy at baseline* and on day 8 and day 15. Tumor biopsy samples are examined by IHC for evaluation of EGFR, phospho-EGFR, HER2, phospho-HER2, phospho-Akt, and phospho-MAPK. Samples are also examined for cell proliferation by Ki-67, apoptosis by TUNEL, and angiogenesis by microvessel density. Additionally, mRNA is extracted from fresh frozen samples and examined by microarray analysis.

NOTE: *Archival tissue acceptable for baseline sample, if available

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer meeting 1 of the following criteria:

  * Locally recurrent disease
  * Locally advanced disease AND meets the following criterion:

    * Chemotherapy-refractory disease (achieved < partial response to ≥ 3 courses of neoadjuvant chemotherapy)
  * Metastatic disease
* Evaluable disease by exam and/or imaging studies

  * Amenable to serial biopsies by skin punch, core biopsy, or fine-needle aspiration
* Unresectable disease after standard neoadjuvant chemotherapy

  * Resectability must be determined by a surgical oncologist prior to treatment
* Stable CNS metastases allowed
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Male or female
* Menopausal status not specified
* Life expectancy > 12 weeks
* ECOG performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow and retain oral medication
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Total bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* Cardiac ejection fraction normal by ECHO or MUGA
* No other malignancy within the past 5 years
* No concurrent disease or condition that would preclude study participation
* No ongoing coagulopathy
* No active severe infection

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy
* At least 3 weeks since prior and no other concurrent systemic therapy for breast cancer
* At least 14 days since prior and no concurrent herbal or alternative medicine
* At least 14 days since prior and no concurrent dietary supplement
* At least 14 days since prior CYP3A4 inducers
* At least 7 days since prior CYP3A4 inhibitors
* No antacid within 1 hour before or after study drug administration
* Concurrent bisphosphonate allowed
* No concurrent oral glucocorticosteroid > 1.5 mg of dexamethasone (or equivalent)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-04; Primary Completion 2010-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Toxicity as assessed by NCI CTCAE v3.0 | 4-5 years
Inhibition of receptor and downstream signal transduction pathway activation in tumor tissue as assessed by IHC | 4-5 years

SECONDARY OUTCOMES:
Efficacy | 4-5 years
Correlation of response with inhibition of downstream signaling | 4-5 years
Gene expression | 4-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C. Dees, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States